CLINICAL TRIAL: NCT01862562
Title: Randomized Controlled Trial to Evaluate Laparoscopic Versus Open Surgery in Elderly Colorectal Cancer Patients Who Were 75 Years Old or Over
Brief Title: Trial to Evaluate Laparoscopic Versus Open Surgery in Elderly Colorectal Cancer Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shoichi Fujii, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Shoichi Fujii, MD, PhD, Associate Professor, Yokohama City University Medical Center
Organization: Yokohama City University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YCUMC-D1108015; YokohamaCUMC34 (Other: YokohamaCUMC)
Record Dates: First submitted 2013-05-16; First posted 2013-05-24 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Colorectal Cancer
Keywords: Laparoscopic surgery; Colorectal cancer; Elderly patient; Randomized control study
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Conversion to Open Surgery; Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open surgery (Active Comparator): Conventional procedure
  Interventions: Procedure: Open surgery
- Laparoscopic surgery (Experimental): Minimum invasive procedure
  Interventions: Procedure: Laparoscopic surgery

INTERVENTIONS:
Procedure: Open surgery — Conventional technique
  Other Names: Open
  Arms: Open surgery
Procedure: Laparoscopic surgery — New minimum invasive technique
  Other Names: Laparoscopic
  Arms: Laparoscopic surgery

SUMMARY:
Elderly patients have poorer preoperative conditions than younger patients. Therefore, minimally invasive surgery should be an effective treatment method for elderly patients. The investigators conducted a randomized trial that compared laparoscopic surgery and conventional open surgery in elderly patients who were 75 years old or over. The purpose of the present study was to clarify the effect of laparoscopic surgery in elderly patients. In our hypothesis of this trial, laparoscopic surgery is superior to conventional open surgery in short-term results, and same outcome in long -term results. Therefore, laparoscopic surgery would be recommended as standard procedure in an elderly colorectal patient.

DETAILED DESCRIPTION:
Patients

* This was a randomized controlled trial conducted at a single institute, which was Yokohama City University Medical Center (Japan).
* 200 patients were age of 75 years old or over were randomly allocated to receive laparoscopic surgery or conventional open surgery.

Surgical procedures

* All surgical procedures were performed by one specialized colorectal treatment team. The laparoscopic surgeries were performed by a surgeon who passed the skill accreditation system for laparoscopic gastroenterological surgery was established by the Japanese Society for Endoscopic Surgery (JSES), and all open surgeries were performed under the supervision of these skillful surgeons.
* All operations were performed according to the standard radical cure procedure described in the seventh edition of the Japanese General Rules for Clinical and Pathological Studies on Cancer of the Colon, Rectum and Anus. That is, intestinal excision with lymph node dissection that separated the feeding blood vessel at its origin was performed in all surgical procedures. Patients who underwent palliative partial excision were not included.
* In the laparoscopic surgery, a medial-to-lateral approach was performed in all patients.
* In the conventional open surgery, the first procedure was done in lateral approach. The reconstruction techniques were the same as those used in laparoscopic surgery.

Randomization

* To balance the operative backgrounds between the laparoscopic and the conventional open surgery groups, the patients were stratified by the tumor location (right colon, left colon and rectum).
* A transverse colon cancer was allocated to the right colon group, and a rectosigmoid cancer was allocated to the rectum group.

Adjuvant therapy

* When the pathological stage was diagnosed as stage 3 by histological examination of the resected specimen, adjuvant chemotherapy was done with oral fluoropyrimidine anti-cancer drug.
* Neither radiation therapy nor preoperative chemotherapy was given to any patient. Preoperative chemo-radiotherapy even for rectal cancer is not yet standard treatment in Japan.

Assessment parameters

* The preoperative parameters
* Operative assessment parameters
* Postoperative assessment parameters An early postoperative complication was defined as a complication that occurred between the finish of the operation and postoperative day 30. A late postoperative complication was defined as a complication that occurred after postoperative day 30. The terminologies of complications were classified according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, and grading was done by Classification of Surgical Complication.
* The pathological results were recorded according to the 7th edition of the Japanese General Rules for Clinical and Pathological Studies on Cancer of the Colon, Rectum and Anus and 7th edition of primary tumor, regional nodes, metastasis (TNM) classification. Circumferential margin involvement was defined as exposure of a cancer cell at the vertical dissection surface on histological examination.
* Quality of life (QOL) scores. The QOL score was measured using the 36-item Short Form Health Survey (SF-36) version 2.0. It is a tool that measures health-related QOL (HRQOL) according to an inclusive standard and not a disease-specific standard. The SF-36 is composed of 36 questions. The score is expressed numerically by the provided scoring algorithm. SF-36 questionnaires were sent to the patients at one month, 6 months and one year after the surgery by postal mail. A return envelope was enclosed with the SF-36 questionnaire, and the patient sent it back to the research secretariat by postal mail. A questionnaire on the defecation situation and wound pain besides the SF-36 was added all three times. The question of when complete rehabilitation occurred was added in the questionnaire at one year.

Follow-up schedule

- The follow-up schedule was as follows according to stage. Patients with stages 0 and 1 were followed up with outpatient examinations including tumor marker measurements, and chest, abdominal and pelvic computed tomography (CT) once a year for five years. Patients with stage 2 and 3a were examined by CT and tumor marker measurements every six months for the first two years. These examinations were done once a year from the third year to the fifth year. Patients with stage 3b and 3c were examined by CT and tumor marker measurements every four months for the first two years, and every six months from the third year to the fifth year.

Statistical analysis

* The primary endpoint was early complication rate.
* The secondary endpoints were 5-year overall survival, 3-year recurrence-free survival, length of postoperative hospital stay, and HRQOL score.
* A sample size of 200 patients was assured to achieve a power of more than 80% to detect a difference between the groups using a two-sided Chi-squared test with type I error rate equal to 0.05, when the true complication rates were 20% and 40% for the laparoscopic and open surgeries, respectively.
* For continuous variables, data are presented as means ± standard deviation (SD). For categorical variables, data are presented as frequencies and percentages (%). Comparison of the endpoints was based on intention-to-treat principle, that is, the patients who switched to another group during surgery were treated as members of the allocated group. The Chi-squared test was applied to evaluate the significance of differences in proportions, and t-test was used to evaluate the significance of differences in continuous variables. A p-value of less than 0.05 was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age of 75 years old or over
* Histologically proven adenocarcinoma
* Clinical tumor penetrates visceral peritoneum (T4a), no metastasis (M0) or lower T factor
* Elective operation
* Tolerable surgery under general anesthesia
* No bulky tumor larger than 8cm in diameter
* No history of laparotomy for colorectal resection except appendectomy
* Provided written informed consent

Exclusion Criteria:

* Synchronous or metachronous (within 5 years) malignancy in another organ except carcinoma in situ
* Multiple colorectal cancer that needs reconstruction two or more times
* Acute intestinal obstruction or perforation due to colorectal cancer
* Lower rectal cancer that required pelvic side wall lymphadenectomy
* Pregnant or lactating women

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-08; Primary Completion 2012-08 (Actual); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Early complication rate | 30 days after surgery
  All complication due to surgical procedure within 30 days after surgery

SECONDARY OUTCOMES:
Overall survival | 5 years
  All death is defined as an event of overall survival. The overall survival rate is appropriate to evaluate whether laparoscopic surgery influences survival which is the true target of malignant disease treatment for curable colorectal cancer by surgery.
Recurrence-free survival | 3 years
  All death and recurrence from colorectal cancer are defined as an event of recurrence-free survival.
Length of postoperative hospital stay | 9 days
  Length of postoperative hospital stay is defined as a duration between surgery and first discharge. An expected average is 9days.
Health-related QOL score | 1 year after surgery
  Short-Form 36 (SF36) is used for measurement of Health-related QOL score. SF-36 questionnaires were sent to the patients at one month, 6 months and one year after the surgery by postal mail. A return envelope was enclosed with the SF-36 questionnaire, and the patient sent it back to the research secretariat by postal mail. A questionnaire on the defecation situation and wound pain besides the SF-36 was added all three times. The question of when complete rehabilitation occurred was added in the questionnaire at one year.

CONTACTS AND LOCATIONS:
Overall Officials: Chikara Kunisaki, Professor, Study Chair — Yokohama City University, Gastroenterological Center
Locations (1):
- Yokohama City University Medical Center, Yokohama, Kanagawa, Japan

REFERENCES:
- [Derived] Ishibe A, Ota M, Fujii S, Suwa Y, Suzuki S, Suwa H, Momiyama M, Watanabe J, Watanabe K, Taguri M, Kunisaki C, Endo I. Midterm follow-up of a randomized trial of open surgery versus laparoscopic surgery in elderly patients with colorectal cancer. Surg Endosc. 2017 Oct;31(10):3890-3897. doi: 10.1007/s00464-017-5418-z. Epub 2017 Feb 15. PMID 28205033